CLINICAL TRIAL: NCT07313072
Title: Topical Use of 2% Tofacitinib for Nail Psoriasis: an Exploratory Clinical Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Principal Investigator, Doris Hexsel, Dr, Hexsel Dermatology Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-DPCHD25-04
Record Dates: First submitted 2025-12-09; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Nail Psoriasis
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medicated Nail Lacquer (Experimental)
  Interventions: Drug: Topical 2% Tofacitinib

INTERVENTIONS:
Drug: Topical 2% Tofacitinib — Each study participant will receive a bottle of nail lacquer containing 2% tofacitinib. Application will be the responsibility of the participant and must be performed once daily throughout the entire study period.

SUMMARY:
To evaluate the efficacy and safety of topical 2% tofacitinib nail lacquer in nail psoriasis, using the NAPSI and DLQI scales before and after 26 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria: Age ≥ 18 years;

* Presence of nail psoriasis in at least one fingernail or toenail;
* Patients not using systemic medication, or without adequate response to systemic medication after at least 6 months of use;
* Ability to read, understand, and sign the Informed Consent Form (ICF) and the Consent Form for Images, Presentations, and Scientific Publications.

Exclusion Criteria: Pregnant or breastfeeding women or those planning to become pregnant during the study period;

* History of sensitivity to any components of the study product;
* Initiation of systemic medication for nail psoriasis less than six months prior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The efficacy of topical 2% tofacitinib | 26 weeks
  The Nail Psoriasis Severity Index (NAPSI) evaluates nail psoriasis severity by assessing a target nail for nail matrix and nail bed involvement. The nail is divided into four quadrants. Nail matrix psoriasis includes pitting, leukonychia, red spots in the lunula, and nail plate crumbling, while nail bed psoriasis comprises onycholysis, splinter hemorrhages, oil drop (salmon patch) discoloration, and nail bed hyperkeratosis. Each component is scored from 0 to 4 according to the number of quadrants affected (1 = 1/4, 2 = 2/4, 3 = 3/4, 4 = 4/4). The total NAPSI score per nail is calculated as the sum of matrix and nail bed scores, ranging from 0 to 8. The score is directly proportional to disease severity, with higher scores indicating greater nail involvement and a score of zero representing absence of nail manifestations. In clinical studies, a decrease in NAPSI score over time indicates clinical improvement.

SECONDARY OUTCOMES:
Safety, Quality of Life, and Treatment Adherence with 2% Tofacitinib | 26 weeks
  The Dermatology Life Quality Index (DLQI) is a validated, standardized instrument used to assess the impact of dermatological diseases on patients' quality of life over the preceding seven days. The questionnaire consists of 10 items covering symptoms and feelings, daily activities, leisure, work or school, personal relationships, and treatment-related burden. Each item is scored on a four-point scale from 0 to 3, where 0 indicates "not at all" and 3 indicates "very much." The total DLQI score is calculated as the sum of all items, yielding a minimum score of 0 and a maximum score of 30. Interpretation is directly proportional to disease impact: higher scores reflect greater impairment and worse dermatology-related quality of life, whereas lower scores indicate less impact, with a score of zero representing no effect on quality of life.

OTHER OUTCOMES:
Monitoring of treatment adherence | 26 weeks.
  This study evaluates the use of a medicated nail lacquer for the treatment of nail psoriasis, and one of the outcome measures will be the monitoring of treatment adherence, including the frequency of application and the correct execution of the nail lacquer application technique. Adherence will be systematically monitored throughout the study period using structured records to verify whether the product is applied in accordance with the dosing regimen and protocol-defined instructions. This monitoring aims to ensure intervention fidelity and to support the accurate interpretation of the treatment's efficacy and safety outcomes.